CLINICAL TRIAL: NCT01035151
Title: Social Ecological Based Smoking Cessation Intervention in Public Housing Neighborhoods
Brief Title: Smoking Cessation Intervention in Public Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUS08022834; R01HL090951 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Cigarette Smoking
Keywords: randomized cluster design; tobacco cessation; smoking cessation; African American
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed Control (Active Comparator): Women in the delayed control condition received culturally sensitive smoking cessation written materials at week 1, and mailed materials at week 6, 12, and 18. At the end of the study (i.e., after the 12 month data collection), participants were offered counseling, nicotine patches, and community health worker contacts.
  Interventions: Behavioral: Control
- Experimental (Experimental): Women in neighborhoods randomized to the S2S received 24-week bundled multi-level intervention. Individual-led strategies were led by paid community health workers (CHWs). The CHWs provided 1:1 contact to reinforce social support, and enhanced self-efficacy with cessation attempts. A certified smoking cessation counselor led behavioral group sessions using the S2S handbook based on the PHS Guidelines. The weekly group sessions were initiated during the 1st week of the intervention, with a total of 6 group sessions over a 6-week period. Transdermal nicotine patches were offered to participants who set a quit date. Within the 24-week study period, the neighborhood tenant association, in partnership with study staff, implemented at least two neighborhood level anti-smoking activities
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — Neighborhood level interventions, peer group (counseling, NRT), and individual level (Coach/CHW)
  Arms: Experimental
Behavioral: Control — Written Cessation Materials
  Arms: Delayed Control

SUMMARY:
The major aim of this study is to test the effectiveness of a bundled, multi-level intervention (Sister to Sister) on smoking cessation outcomes in female smokers residing in public housing neighborhoods.

Hypothesis 1.1: As compared to the control group, women receiving the Sister to Sister Intervention will have higher 7-day point prevalence quit rates at 6- and 12-months as validated by salivary cotinine.

Hypothesis 1.2: As compared to the control group, women receiving the Sister to Sister Intervention will have higher 6- and 12-month prolonged smoking abstinence as validated by salivary cotinine.

DETAILED DESCRIPTION:
This was a cluster randomized controlled study evaluating the effect of a multi-level intervention, Sister to Sister, on the smoking cessation in two Southeastern US metropolitan areas. Fourteen subsidized housing neighborhoods, eight in Charleston, SC and six in Augusta, GA, were pair matched based on size; with one neighborhood in each pair randomized to the intervention to ensure balanced recruitment between groups. Neighborhoods ranged in size from 22 to 33 participants with a total sample size of 409 women; neighborhoods were chosen as the primary sampling unit to prevent contamination of the outcome within neighborhoods, with women in the neighborhoods as secondary sampling unit. All statistical analyses were conducted using SAS 9.2 (SAS Institute, Cary, NC) with statistical significance at an alpha level of 0.05. Comparison between groups at baseline used t-tests for continuous variables and chi-square tests for categorical variables. The primary outcome of interest was smoking status which was dichotomized (smoker/non-smoker) at the 6 and 12 month measurements. Smoking status was determined by cotinine levels in saliva with non-smokers defined as those with cotinine levels of 14 ng/mL or less.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age and older,
* female, resident of public housing, daily smoker

Exclusion Criteria:

* pregnant,
* breastfeeding,
* no intentions to quit smoking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-07; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Andrews, PhD, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Medical College of Georgia, Augusta, Georgia
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Contact the PI

REFERENCES:
- [Background] Andrews JO, Mueller M, Newman SD, Magwood G, Ahluwalia JS, White K, Tingen MS. The association of individual and neighborhood social cohesion, stressors, and crime on smoking status among African-American women in southeastern US subsidized housing neighborhoods. J Urban Health. 2014 Dec;91(6):1158-74. doi: 10.1007/s11524-014-9911-6. PMID 25316192
- [Background] Spruill IJ, Leite RS, Fernandes JK, Kamen DL, Ford ME, Jenkins C, Hunt KJ, Andrews JO. Successes, Challenges and Lessons Learned: Community-engaged research with South Carolina's Gullah population. Gateways. 2013;6:10.5130/ijcre.v6i1.2805. doi: 10.5130/ijcre.v6i1.2805. No abstract available. PMID 25364473
- [Background] Andrews JO, Newman SD, Heath J, Williams LB, Tingen MS. Community-based participatory research and smoking cessation interventions: a review of the evidence. Nurs Clin North Am. 2012 Mar;47(1):81-96. doi: 10.1016/j.cnur.2011.10.013. Epub 2011 Dec 14. PMID 22289400
- [Background] Andrews JO, Tingen MS, Jarriel SC, Caleb M, Simmons A, Brunson J, Mueller M, Ahluwalia JS, Newman SD, Cox MJ, Magwood G, Hurman C. Application of a CBPR framework to inform a multi-level tobacco cessation intervention in public housing neighborhoods. Am J Community Psychol. 2012 Sep;50(1-2):129-40. doi: 10.1007/s10464-011-9482-6. PMID 22124619
- [Background] Magwood GS, Andrews JO, Zapka J, Cox MJ, Newman S, Stuart GW. Institutionalization of community partnerships: the challenge for academic health centers. J Health Care Poor Underserved. 2012 Nov;23(4):1512-26. doi: 10.1353/hpu.2012.0161. PMID 23698666
- [Background] Newman SD, Andrews JO, Magwood GS, Jenkins C, Cox MJ, Williamson DC. Community advisory boards in community-based participatory research: a synthesis of best processes. Prev Chronic Dis. 2011 May;8(3):A70. Epub 2011 Apr 15. PMID 21477510
- [Result] Andrews JO, Mueller M, Dooley M, Newman SD, Magwood GS, Tingen MS. Effect of a smoking cessation intervention for women in subsidized neighborhoods: A randomized controlled trial. Prev Med. 2016 Sep;90:170-6. doi: 10.1016/j.ypmed.2016.07.008. Epub 2016 Jul 14. PMID 27423320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 34 subsidized housing neighborhoods in these two regions, the study was implemented in the 14 neighborhoods that met eligibility. Seven matched pairs were formed and randomly assigned one neighborhood in each pair to either the treatment condition or a delayed control condition. 27-32 participants enrolled in each neighborhood.
Pre-assignment Details: Common reasons for exclusions were not a resident of the neighborhood, not an active smokers.
Period: Overall Study
Arm/Group | Delayed Control | Experimental
Started | 209 | 200
Completed | 188 | 185
Not Completed | 21 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Control | Experimental | Total
Number analyzed (Participants) | 209 | 200 | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15.6) | 41 (14.1) | 42 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 200 | 409
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 190 | 180 | 370
  Unknown or Not Reported | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 192 | 157 | 349
  White | 11 | 28 | 39
  More than one race | 2 | 13 | 15
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 209 | 200 | 409
Nicotine Dependence Score [Mean (Standard Deviation); unit: units on a scale] — The Fagerstrom Test for Nicotine Dependence was assessed to measure nicotine dependence. The scale ranges from minimum score of 0 to a maximum score of 10. The higher the score, the higher the nicotine dependence.
  units on a scale | 4.8 (2.2) | 4.7 (2.2) | 4.7 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Abstinent From Smoking
Description: Reported abstinence validated by exhaled CO and saliva cotinine
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Control | Experimental
Number analyzed (Participants) | 188 | 185
Participants | 10 | 24

ADVERSE EVENTS:
Time Frame: 12 month study period
Description: Collected data on self reported serious adverse events from nicotine patch use, behavioral counseling
Arm/Group | Delayed Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/209 | 0/200
Other Adverse Events (participants affected / at risk) | 0/209 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT01035151/SAP_000.pdf
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT01035151/Prot_001.pdf